CLINICAL TRIAL: NCT07407933
Title: A Phase Ib/II, Multicenter, Open-Label Study to Evaluate Safety, Efficacy, and Pharmacokinetics of YL201 in Combination With Other Anti-Cancer Therapies in Patients With Advanced Solid Tumors
Brief Title: A Study of YL201 in Combination With Other Anti-Cancer Therapies in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL201-INT-102-02
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Thoracic Neoplasms, Lung Diseases, Small Cell Lung Carcinoma
Keywords: Small cell lung cancer, Antibody drug conjugate, YL201, atezolizumab
MeSH Terms: conditions — Thoracic Neoplasms; Lung Diseases; Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- YL201 1.2mg/kg in combination with atezolizumab 1200mg Q3W (Experimental)
  Interventions: Drug: YL201; Drug: Atezolizumab
- YL201 1.6mg/kg in combination with atezolizumab 1200mg Q3W (Experimental)
  Interventions: Drug: YL201; Drug: Atezolizumab
- YL201 2.0mg/kg in combination with atezolizumab 1200mg Q3W (Experimental)
  Interventions: Drug: YL201; Drug: Atezolizumab

INTERVENTIONS:
Drug: YL201 — YL201 intravenous infusion will be administered on Day 1 of each 21-day cycle.
Drug: Atezolizumab — Atezolizumab intravenous infusion will be administered at a dose of 1200 mg on Day 1 of each 21-day cycle

SUMMARY:
This is a phase Ib/II, multicenter, open-label study of YL201 combined with atezolizumab. The study will include 2 parts. Part 1 of the study is a dose escalation in participants with previously untreated ES-SCLC to determine the safety and tolerability of YL201 in combination with fixed dose of atezolizumab. The planned dose levels of YL201 are 1.2 mg/kg, 1.6 mg/kg and 2.0 mg/kg. Part 2 consists of a dose optimization stage followed by a dose expansion stage. During the dose optimization stage, participants will be randomized 1:1:1 to receive either YL201 at 1.2 mg/kg,1.6 mg/kg or 2.0 mg/kg Q3W in combination with fixed dose of atezolizumab. The decision to initiate the dose expansion stage in Part 2 and choose one or two of the YL201 dose level(s) will be based on the review of safety, PK, and efficacy from the dose optimization stage. Treatment will continue until disease progression, unacceptable toxicity, or withdraw of consent.

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age or older. 2. Histologically or cytologically confirmed diagnosis of ES-SCLC 3. Eastern Cooperative Oncology Group performance status of 0 or 1 4. Adequate hematologic and end-organ function

Exclusion Criteria:

1. No prior systemic anti-cancer treatment for ES-SCLC
2. No prior treatment targeting B7H3 or topoisomerase I inhibitor
3. No clinically active brain metastases or spinal cord compression
4. No current or history of interstitial lung disease (ILD)/ pneumonitis
5. No clinically significant cardiovascular disease (eg, New York Heart Association class II to IV congestive heart failure)

Other protocol-defined inclusion/ exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Nature and Frequency with Dose-Limiting Toxicities (DLTs) | 21 days
Adverse Events | First dose of study treatment up to disease progression or death from any cause (up to approximately 6 years)
  Incidence, nature, and severity of AEs graded according to the NCI CTCAE v5

SECONDARY OUTCOMES:
ORR | Up to approximately 3 years
DOR | Up to approximately 3 years
PFS | Up to approximately 3 years
OS | Up to approximately 3 years
AUC | Up to approximately 3 years
CL | Up to approximately 3 years
Vss | Up to approximately 3 years
t1/2 | Up to approximately 3 years
Cmax | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No